CLINICAL TRIAL: NCT03734588
Title: Dose-finding Study of SPK-8016 Gene Therapy in Patients With Hemophilia A to Support Evaluation in Individuals With FVIII Inhibitors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPK-8016-101
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Adeno-Associated Virus (AAV); Blood Coagulation Disorder; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Factor VIII (FVIII); Factor VIII (FVIII) Deficiency; Factor VIII (FVIII) Gene; Factor VIII (FVIII) Protein; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Gene Therapy; Gene Transfer; Hematologic Diseases; Hemorrhagic Disorders; Recombinant; Vector; Inhibitors
MeSH Terms: conditions — Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemophilia A; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hematologic Diseases; Hemorrhagic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPK-8016 (Experimental): All participants who meet the eligibility criteria will receive an outpatient single intravenous (i.v.) administration of SPK-8016.
  Interventions: Genetic: SPK-8016

INTERVENTIONS:
Genetic: SPK-8016 — adeno-associated viral vector

SUMMARY:
SPK-8016 is in development for the treatment of patients with inhibitors to FVIII. This Phase 1/2, open-label, non-randomized, dose-finding study to evaluate the safety, efficacy, and tolerability of SPK-8016 in adult males with severe hemophilia A and no measurable inhibitor against FVIII.

ELIGIBILITY:
Inclusion Criteria:

1. Be male and ≥18 years of age;
2. Have clinically severe hemophilia A, defined as:

   1. <1% (<1 IU/dL) endogenous FVIII activity levels as historically documented by a certified laboratory or screening data results; OR
   2. 1-2% (1-2 IU/dL) endogenous FVIII activity levels and > 10 bleeding events per year (in the last 52 weeks prior to screening); OR
   3. 1-2% (1-2 IU/dL) endogenous FVIII activity levels and on prophylaxis;
3. Have had >150 exposure days (EDs) to any recombinant and/or plasma-derived FVIII concentrates or cryoprecipitates
4. Have no prior history of hypersensitivity or anaphylaxis associated with any FVIII or IV immunoglobulin administration
5. Have no measurable inhibitor against FVIII as assessed by central laboratory, have no confirmed history of clinically significant FVIII inhibitor, and no clinical signs or symptoms of decreased response to FVIII administration (Note: family history of inhibitors will not exclude study participation)
6. Agree to use reliable barrier contraception after the administration of SPK-8016 until notified by the Investigator.

Exclusion Criteria:

1. Have active hepatitis B or C
2. Have significant underlying liver disease.
3. Have serological evidence of HIV-1 or HIV-2 with CD4 counts ≤200/mm3. Participants who are HIV-positive and stable, with an adequate CD4 count (>200/mm3) and undetectable viral load, and are on an antiretroviral drug regimen are eligible to enroll
4. Have detectable antibodies reactive with AAV-Spark capsid
5. Have history of chronic infection or other chronic disease
6. Have been dosed in a previous gene therapy research trial within the last 52 weeks or with an investigational drug within the last 12 weeks
7. Any concurrent clinically significant major disease (such as liver abnormalities or type I diabetes) or other condition that, in the opinion of the Investigator and/or Sponsor, makes the subject unsuitable for participation in the study;
8. Unable or unwilling to comply with the schedule of visits and study assessments described in the clinical protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetically male
Enrollment: 4 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Chang, MD, Study Director — Spark Therapeutics, Inc.
Locations (11):
- United States (11):
  - Orthopaedic Institute for Children, Los Angeles, California
  - Illinois Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Weill Cornell Medicine, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A dose-finding part of this trial was planned but no participants were enrolled into the higher dose arms. All participants received SPK-8016 5x10^11 vg/kg
Groups:
- SPK-8016: Participants received a single intravenous infusion of SPK-8016 at 5x10^11 vector genomes per kilogram body weight (vg/kg).
Period: Overall Study
Arm/Group | SPK-8016
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all enrolled participants who received the infusion of SPK-8016.
Groups:
- SPK-8016: Participants received a single intravenous infusion of SPK-8016 at 5x10^11 vg/kg.
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (19.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Participants With Hepatic Transaminase Elevation Requiring Immunosuppression.
Time Frame: Up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Peak FVIII Activity Levels Assessed by Coagulation Clotting Assays
Time Frame: Up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Number; unit: percentage of normal activity
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
percentage of normal activity | NA — Data was not analyzed due to low number of participants enrolled. Data values are not reported due to privacy concerns related to low enrollment.

4. Primary Outcome: Steady-state FVIII Activity Levels Assessed by Coagulation Clotting Assays
Time Frame: Up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Mean (Standard Deviation); unit: percentage of normal activity
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
percentage of normal activity | NA (NA) — Insufficient number of participants with events

5. Primary Outcome: Number of Bleeding Events (Spontaneous and Traumatic) Since 28 Day Post Vector Administration
Time Frame: From 28 days post vector administration up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Number; unit: Number of bleeding events
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Number of bleeding events
  Traumatic | 6
  Spontaneous | 1

6. Primary Outcome: Annualized Infusion Rate
Time Frame: From 28 days post vector administration up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Number; unit: Annualized Infusion Rate
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Annualized Infusion Rate | NA — Data was not analyzed due to low number of participants enrolled. Data values are not reported due to privacy concerns related to low enrollment.

7. Secondary Outcome: Time to Achieve Steady-state FVIII Activity Levels
Time Frame: Up to week 52
Population: The FAS included all enrolled participants who received the infusion of SPK-8016.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
hours | NA (NA) — Insufficient number of participants with events

8. Secondary Outcome: Number of Participants With Vector-shedding of SPK-8016 in Bodily Fluids
Time Frame: Up to week 52
Population: Results were uninterpretable due to a technical error.
Arm/Group | SPK-8016
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Immune Responses to AAV Capsid Protein and BDD-hFVIII Transgene
Time Frame: Up to week 52
Population: The FAS includes all enrolled participants who received the infusion of SPK-8016.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8016
Number analyzed (Participants) | 4
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to week 52
Arm/Group | SPK-8016
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPK-8016 (N=4)
Food Poisoning (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPK-8016 (N=4)
Cushingoid (Endocrine disorders) | 1
Vision Blurred (Eye disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tooth Loss (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Feeling Hot (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Swelling Face (General disorders) | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1
Candida Infection (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Limb Crushing Injury (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Blood Glucose Increased (Investigations) | 1
Weight Increased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Joint Noise (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Libido Decreased (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03734588/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03734588/SAP_001.pdf